CLINICAL TRIAL: NCT03122769
Title: Cardiac Uptake of Metformin and Expression of Metformin Membrane Transporter Proteins in the Human Failing Myocardium
Brief Title: Cardiac Uptake of Metformin, Visualized by Positron Emission Tomography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henrik Wiggers (Other)
Responsible Party: Sponsor-Investigator, Henrik Wiggers, Senior consultant, associate professor, MD, PhD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-003453-15
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure, Systolic
Keywords: Metformin; Heart Failure; Organic cation transporter; Pharmacogenetics; Pharmacokinetics; Positron Emission Tomography
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: All 6 subjects allocated to the study will receive 11C-metformin intravenously.
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 11C-metformin (Experimental): All participants allocated to the study will be included in this arm
  Interventions: Radiation: 11C-metformin

INTERVENTIONS:
Radiation: 11C-metformin — 200 MBq of 11C-metformin is injected in the cubital vein. The participant is then scanned for 120 min using Positron Emission Tomography

SUMMARY:
The purpose of the study is to evaluate if metformin is taken up into the failing myocardium. Recent experimental and epidemiological studies have shown beneficial effects of metformin on heart failure. It is unknown whether this effect is direct or indirect.

The aim of the study is to investigate if metformin is taken up in heart failure using a novel 11C-metformin tracer and positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure, Left Ventricular Ejection Fraction <45%
* New York Heart Association (NYHA) class I, II, III
* Relatively preserved renal function (eGFR > 30 ml/min)
* Ability to understand the written patient information and to give informed consent
* Negative p-HCG for women of childbearing potential

Exclusion Criteria:

* Known allergy to metformin
* Age < 18 years
* Current abuse of alcohol or drugs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Metformin uptake in the failing myocardium | 12 months
  Cardiac uptake is evaluated through analysis of acquired PET-images.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark